CLINICAL TRIAL: NCT01649570
Title: An Open-labelled, Single-arm, Multi-centre, 6-month Study to Investigate the Safety and Efficacy of NovoRapid as Meal Time Insulin in Type 2 Diabetes Patients Treated on a Basal-bolus Regimen With NPH Human Insulin
Brief Title: Safety and Efficacy of Insulin Aspart in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Public Access to Clinical Trials, Novo Nordisk A/S
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1472
Record Dates: First submitted 2011-11-25; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin aspart (Experimental)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Administrated subcutaneously (s.c., under the skin) three times a day before each meal for 24 weeks

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the safety and efficacy of NovoRapid® (insulin aspart) as meal time insulin in subjects with type 2 diabetes treated on a basal-bolus regimen with Neutral Protamine Hagedorn (NPH) human insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treated with insulin for at least 12 months and currently on a basal-bolus regimen for at least 12 weeks
* HbA1c below or equal to 11.0%
* BMI (body mass index) below 30 kg/m^2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2002-03; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoglycaemia

SECONDARY OUTCOMES:
Incidence of adverse events (AEs)
Clinical laboratory tests: Haematology and biochemistry
Insulin antibodies
Glycaemic control parameters: Glycosylated haemoglobin A1c (HbA1c), fasting plasma glucose (FPG) and post-prandial plasma glucose (PPPG)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com